CLINICAL TRIAL: NCT05118724
Title: Perioperative/Adjuvant Atezolizumab in Patients With MSI-high or MMR-deficient Stage II High Risk and Stage III Colorectal Cancer Ineligible for Oxaliplatin-based Chemotherapy - a Phase II Study
Brief Title: Atezolizumab in Patients With MSI-h/MMR-D Stage II High Risk and Stage III Colorectal Cancer Ineligible for Oxaliplatin
Acronym: ANTONIO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Roche Pharma AG (Industry); Immodulon Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-KRK-0220
Record Dates: First submitted 2021-10-08; First posted 2021-11-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: MSI-high; MMR-deficient; Stage III Colorectal Cancer; stage II high risk Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Turcot syndrome | interventions — atezolizumab; IMM-101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atezolizumab (Experimental): Atezolizumab 840mg i.v. (q2w) for a total of 12 cycles (24 doses)
  Interventions: Drug: Atezolizumab
- IMM-101 plus atezolizumab (Experimental): One initial dose of IMM-101 intradermally at 1.0 mg 14 ±2 days before start of atezolizumab treatment (same as Arm A)
  Interventions: Drug: Atezolizumab; Drug: IMM-101

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 840mg i.v., on Day 1 and Day 15 (q2w) of every 28-day treatment cycle for a total of 12 cycles (24 doses)
  Other Names: Tecentriq
Drug: IMM-101 — Suspension of Heat-Killed Whole Cell Mycobacterium obuense (NCTC 13365) in Borate Buffered Saline for Intradermal Injection
  Arms: IMM-101 plus atezolizumab

SUMMARY:
The investigators hypothesize that atezolizumab will improve the prognosis of patients with stage III dMMR CRC ineligible for or refusing oxaliplatin-based adjuvant chemotherapy compared to SOC and that these could therefore be promising therapeutic options.

DETAILED DESCRIPTION:
The current standard of care for adjuvant treatment of oxaliplatin-ineligible patients with stage III dMMR colon cancer is fluoropyrimidine monotherapy. In the COLOPREDICT registry, the 3 years DFS rate for such patients >70 years of age is 63% (95%CI: 53-75%). In contrast to patients with mismatch repair proficient (pMMR) colon cancer, however, it is not established whether patients with stage III dMMR colon cancer benefit from adjuvant fluoropyrimidine monotherapy at all. For patients with stage II colon cancer in an otherwise identical setting, there is no indication for adjuvant treatment due to a lack of clinical benefit compared to surgery alone. Clinical results suggests a similar situation for stage III malignancy. Siwemilar to other checkpoint inhibitors (CPI), the PD-L1 antibody atezolizumab demonstrated impressive activity and good tolerability in patients with metastatic dMMR CRC. Recently, the randomized phase III Keynote-177 trial was presented. In Keynote-177, patients with dMMR metastatic CRC were randomized to the PD-1 antibody pembrolizumab or to chemotherapy (mFOLFOX6 or FOLFIRI with or without bevacizumab or cetuximab as per Investigator's choice). Pembrolizumab treatment resulted in a statistically significant prolongation of Progression-free survival . In addition, side effects were lower with pembrolizumab and quality of life was improved compared to conventional chemotherapy. Thus, pembrolizumab will become the new standard of care in patients with dMMR metastatic CRC in first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent including participation in translational research and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Male or female ≥ 18 years of age
3. Histologically confirmed adenocarcinoma of the colon or rectum
4. For the main study: Pathological Stage III disease For the perioperative sub-study: Clinical stage III disease
5. For the main study: R0-resected primary tumor For the perioperative sub-study: Resectable primary tumor; R0 resection anticipated (R1-resected patients can remain on study.)
6. Tumor is MSI-high (MSI-H) or MMR-deficient (dMMR) For the main study: assessed from biopsy or from resected tumor tissue For the perioperative sub-study: assessed from biopsy
7. ECOG status 0 - 2
8. Ineligible for oxaliplatin-based adjuvant chemotherapy or patient's refusal of oxaliplatin-based adjuvant chemotherapy. Oxaliplatin ineligibility criteria are:

   * Age ≥70
   * Peripheral sensory neuropathy > grade 1
   * QT interval prolongation or co-medication with drugs known to prolong the QT interval
   * Renal impairment (glomerular filtration rate <60ml per min)
   * Suboptimal controlled diabetes mellitus (HbA1C>6,5%) with the risk of aggravation upon corticoid premedication for oxaliplatin based chemotherapy
9. Adequate blood count, liver enzymes, and renal function - re-testing can be undergone once in case of initial results near cutoff

   * White blood cell count ≥ 3.5 x 106/mL
   * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   * Hemoglobin ≥ 9 g/dL (blood transfusion > 2 weeks before testing is permitted)
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal
   * Serum Creatinine ≤ 1.5 x institutional ULN and a calculated glomerular filtration rate ≥ 30 mL per minute
10. Patients not receiving therapeutic anticoagulation must have an INR < 1.5 ULN and PTT < 1.5 ULN within 7 days prior to registration. The use of full dose anticoagulants is allowed as long as the INR or PTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least three weeks at the time of registration
11. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
12. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly-effective contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) and to continue its use for up to 6 months after the last dose of study drug.

Exclusion Criteria:

1. Severe infection within 4 weeks prior to registration, including, but not limited to, hospitalization for complications of infection, bacteremia, known active pulmonary disease with hypoxia, or severe pneumonia or any active infection (bacterial, viral or fungal) requiring systemic therapy within 4 weeks prior to registration. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.

   Patients with positive test result for SARS-CoV2 should be managed as per local institutional guidelines.
2. For the main study: Distant metastases or residual disease For the perioperative sub-study: Distant metastases or macroscopic residual disease (R2 resection status)
3. Neoadjuvant radiotherapy or radio-chemotherapy (enrollment of rectal cancer patients without prior radio- or radio-chemotherapy is allowed); prior neoadjuvant radio-chemotherapy (RCT) or radiotherapy (RT) for rectal cancer is allowed if >5 years and secondary colorectal cancer
4. Prior adjuvant chemotherapy for colorectal cancer; allowed if >5 years and secondary colorectal cancer
5. Prior treatment with atezolizumab or any other checkpoint inhibitor (anti-PD-1, anti-PD-L1, anti- CTLA-4)
6. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to treatment start, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions: Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible. Inhaled corticosteroids for chronic obstructive pulmonary disease or bronchial asthma, supplemental mineralo-corticosteroids or low-dose corticosteroids for adrenal-cortical insufficiency are allowed
7. Clinically significant cardiovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) 6 months before enrollment.
8. History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins.
9. Known hypersensitivity to CHO cell products or any component of the atezolizumab formulation.
10. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), druginduced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. If any of these lung diseases is suspected based on the patient's history or the integrated evaluation of clinical and radiological records, an additional spirometry should be conducted.
11. Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test at screening. Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test at screening followed by a negative HBV DNA test, are eligible for the study. The HBV DNA test will be performed only for patients who have a positive total HBcAb test. Patients are also eligible if HBV DNA < 500 IU/mL obtained within 28 days prior to initiation of study treatment, AND anti-HBV treatment (per local standard of care; e.g., entecavir) for a minimum of 14 days prior to study entry and willingness to continue treatment for the length of the study.
12. Anti-viral therapy against HCV during the trial (but allowed prior to trial)
13. Positive human immunodeficiency virus (HIV) test. As an exception, known HIV+ patients may be included if they have:

    * A stable regimen of highly active anti-retroviral therapy (HAART)
    * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
    * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based tests
14. a) Treatment with a live, attenuated vaccine within 4 weeks prior to first dose of study treatment, or anticipation of need for such a vaccine during study treatment or within 5 months after the last dose of study treatment. b) Treatment with any vaccine during screening and the first cycle of treatment.
15. Active tuberculosis (as ruled out by clinical evaluation including medical history, physical examination, radiographic findings on baseline CT/ MRI of chest/abdomen/pelvis; if active tuberculosis is suspected, tuberculosis testing should be performed as per local standard of care).
16. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis. The following exceptions apply:

    * Patients with a history of autoimmune-mediated hypothyroidism who are on thyroid replacement hormone are eligible for the study.
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (i.e., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or highpotency or oral corticosteroids within the previous 12 months
17. Prior (<3 years) or concurrent malignancy that either progresses or requires active treatment.

    Exceptions are: basal cell cancer of the skin, pre-invasive cancer of the cervix, T1a or T1b prostate carcinoma, or superficial urinary bladder tumor [Ta, Tis and T1]
18. History of hypersensitivity to any of the study drugs
19. History of allergic reaction to any mycobacterial product
20. Prior allogeneic stem cell or solid organ transplantation requiring immunosuppressive therapy or other major immunosuppressive therapy
21. Severe non-healing wounds, ulcers or bone fractions
22. Evidence of bleeding diathesis or coagulopathy
23. Major gastrointestinal bleeding within 4 weeks prior to treatment start, unless cause of bleeding was the resected tumor
24. Major surgical procedures other than primary tumor resection, except open biopsy, nor significant traumatic injury within 28 days prior to registration, or anticipation of the need for major surgical procedure during the course of the study except for surgery of central intravenous line placement for chemotherapy administration
25. Medication that is known to interfere with any of the agents applied in the trial
26. Female subjects who are pregnant or breast-feeding; male or female patients of reproductive potential who are not employing an effective method of birth control as listed in the protocol (failure rate of less than 1% per year, see protocol section 7.1.3). Women of childbearing potential must have a negative pregnancy test
27. Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or affect patient safety or study results
28. Participation in another clinical study with an investigational drug within 28 days prior to treatment start or 7 half-lives of previously used trial medication, whichever is longer
29. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities (AMG § 40, Abs. 1 No. 4)
30. Affected persons who might be dependent on the sponsor or the investigator

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | at 3 years
  DFS-rate

SECONDARY OUTCOMES:
Disease-free Survival (DFS) | at 1, 2, 5 years
  DFS-rate
Overall Survival (OS) | at 1, 2, 3, 5 years
  OS-rate

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kasper-Virchow, MD, Principal Investigator — Universitätsklinikum Essen
Locations (1):
- Westdeutsches Tumorzentrum, Essen, Germany

IPD SHARING:
Plan to Share IPD: No